CLINICAL TRIAL: NCT04814420
Title: Atrial Fibrosis in Obstructive Sleep Apnea Patients: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-2081
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation; Obstructive Sleep Apnea
Keywords: Ablation; Atrial Fibrosis; Delayed Enhancement Magnetic Resonance Imaging; Electrocardiogram
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Sixty participants would be an adequate sample size for this pilot study to represent all stages of OSA and controls (10 mild, 10 moderate,10 severe OSA with no atrial fibrillation, 10 controls with no OSA and no atrial fibrillation, 10 mild and 10 severe OSA with atrial fibrillation).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Group A (Experimental): Mild OSA
  * 10 patients diagnosed with mild OSA (5<AHI<15) with no atrial fibrillation.
  * Diagnosis confirmed through polysomnography* before enrollment.
  Interventions: Device: Delayed enhancement magnetic resonance imaging (DE-MRI)
- Group B (Experimental): Moderate OSA
  * 10 patients diagnosed with moderate OSA (15<AHI<30) with no atrial fibrillation.
  * Diagnosis confirmed through polysomnography* before enrollment.
  Interventions: Device: Delayed enhancement magnetic resonance imaging (DE-MRI)
- Group C (Experimental): Severe OSA
  * 10 patients diagnosed with severe OSA (AHI>30) with no atrial fibrillation.
  * Diagnosis confirmed through polysomnography* before enrollment.
  Interventions: Device: Delayed enhancement magnetic resonance imaging (DE-MRI)
- Group D (Experimental): Mild OSA and AF
  * At least 10 patients diagnosed with mild OSA (5<AHI<15).
  * Diagnosis confirmed through polysomnography* before enrollment.
  * Diagnosed with AF.
  Interventions: Device: Delayed enhancement magnetic resonance imaging (DE-MRI)
- Group E (Experimental): Severe OSA and AF
  * At least 10 patients diagnosed with severe OSA (AHI>30).
  * Diagnosis confirmed through polysomnography* before enrollment.
  * Diagnosed with AF.
  Interventions: Device: Delayed enhancement magnetic resonance imaging (DE-MRI)
- Group F (Other): Control - No OSA
  10 control patients without OSA and without AF.
  Interventions: Device: Delayed enhancement magnetic resonance imaging (DE-MRI)

INTERVENTIONS:
Device: Delayed enhancement magnetic resonance imaging (DE-MRI) — The patient will be injected with late gadolinium enhancement (0.01 mmol/kg standard dosage), which is a contrast agent used in clinical practice in MRI imaging studies. The contrast agent is used to enhance specific regions/tissues on MRI and, in this study, will allow the investigators to identify fibrotic tissue within the heart. The patient then undergoes the MRI sequence, which lasts approximately 20-25 minutes. Images will be reviewed for quality by trained technicians. This will be repeated after 6 months.

SUMMARY:
The investigators hypothesize that Obstructive Sleep Apnea (OSA) is an independent risk factor for atrial fibrosis development. The investigators aim to prove the presence of atrial fibrosis on Delayed Enhancement Magnetic Resonance Imaging (DE-MRI) in OSA patients without atrial fibrillation (AF).

DETAILED DESCRIPTION:
This is a cross sectional pilot study. Sixty mild to severe OSA patients and five age- and Body Mass Index (BMI)-matched controls will undergo a DE-MRI. Demographics, medical history and polysomnography results will be collected. Patients diagnosed with obstructive sleep apnea have undergone a polysomnography before the study and were diagnosed based on this test. The investigators will not be performing a polysomnography for any of the patients, just collecting the previous results from their medical charts to confirm they have a true OSA diagnosis for their inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

Group A: 10 patients 18-75-year-old With mild OSA (5<AHI<15), confirmed by polysomnography. No previous AF diagnosis on the medical chart

Group B: 10 patients 18-75-year-old With moderate OSA (15<AHI<30), confirmed by polysomnography. No previous AF diagnosis on the medical chart

Group C: 10 patients 18-75-year-old With severe OSA (AHI>30), confirmed by polysomnography. No previous AF diagnosis on the medical chart

Group D (mild OSA+ AF): 10 patients 18-75-year-old With mild OSA (5<AHI<15), confirmed by polysomnography. Previous AF diagnosis

* In this group, patients with AF and OSA who already have done MRI might be included.

Group E (severe OSA +AF): 10 patients 18-75-year-old With severe OSA (AHI>30), confirmed by polysomnography. Previous AF diagnosis

*In this group, patients with AF and OSA who already have done MRI might be included.

Group F (Control): 10 Patients 18-75-year-old No previous OSA and/or AF Diagnosis on the medical chart

Exclusion Criteria:

* History of chronic heart failure (LVEF < 50%), AF, myocardial infarction, valvular disease.
* Prior cardiac or chest surgery.
* Other advanced pulmonary disease (severe Chronic Obstructive Pulmonary Disease (COPD) or asthma, pulmonary hypertension) or central sleep apnea.
* Contraindications to DE-MRI (e.g. allergy to gadolinium, pacemakers, defibrillators (ICD's), other devices/implants contraindicated for MRI, glomerular filtration rate <30 ml/min, etc.).
* Pregnancy.
* Inability to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of atrial fibrosis in the left atrium measured by DE-MRI | Baseline visit
  DE-MRI purpose is to quantify the degree of atrial structural remodeling or fibrosis Left Atrial Volume Max on MRI measurement reflects atrial load to provide insight into atrial remodeling Left Atrial Volume Min on MRI is important for understanding atrial function, particularly its ability to contract and expel blood into left ventricle Left Atrial Volume Index on MRI is an indicator of left atrial enlargement compared to raw volume measurements Left Atrial Emptying Fraction on MRI is a measure of atrial contractile function. Higher LAEF indicates better atrial function, while lower values can signal impaired atrial mechanics Left Atrial Global Strain on MRI which is the percentage change in myocardial length along the long axis of the left atrium, is calculated using a formula averaging the individual longitudinal strain values from each segment of the myocardium, providing a comprehensive measure of myocardial deformation

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Pandey, MD, Principal Investigator — Tulane University Medical Center
Locations (2):
- United States (2):
  - East Jefferson General Hospital, New Orleans, Louisiana
  - Tulane University Medical Center, New Orleans, Louisiana

REFERENCES:
- [Background] May AM, Van Wagoner DR, Mehra R. OSA and Cardiac Arrhythmogenesis: Mechanistic Insights. Chest. 2017 Jan;151(1):225-241. doi: 10.1016/j.chest.2016.09.014. Epub 2016 Sep 29. PMID 27693594
- [Background] Gami AS, Hodge DO, Herges RM, Olson EJ, Nykodym J, Kara T, Somers VK. Obstructive sleep apnea, obesity, and the risk of incident atrial fibrillation. J Am Coll Cardiol. 2007 Feb 6;49(5):565-71. doi: 10.1016/j.jacc.2006.08.060. Epub 2007 Jan 22. PMID 17276180
- [Background] Gami AS, Pressman G, Caples SM, Kanagala R, Gard JJ, Davison DE, Malouf JF, Ammash NM, Friedman PA, Somers VK. Association of atrial fibrillation and obstructive sleep apnea. Circulation. 2004 Jul 27;110(4):364-7. doi: 10.1161/01.CIR.0000136587.68725.8E. Epub 2004 Jul 12. PMID 15249509
- [Background] Kanagala R, Murali NS, Friedman PA, Ammash NM, Gersh BJ, Ballman KV, Shamsuzzaman AS, Somers VK. Obstructive sleep apnea and the recurrence of atrial fibrillation. Circulation. 2003 May 27;107(20):2589-94. doi: 10.1161/01.CIR.0000068337.25994.21. Epub 2003 May 12. PMID 12743002
- [Background] Ng CY, Liu T, Shehata M, Stevens S, Chugh SS, Wang X. Meta-analysis of obstructive sleep apnea as predictor of atrial fibrillation recurrence after catheter ablation. Am J Cardiol. 2011 Jul 1;108(1):47-51. doi: 10.1016/j.amjcard.2011.02.343. Epub 2011 Apr 29. PMID 21529734
- [Background] Linz D, Brooks AG, Elliott AD, Nalliah CJ, Hendriks JML, Middeldorp ME, Gallagher C, Mahajan R, Kalman JM, McEvoy RD, Lau DH, Sanders P. Variability of Sleep Apnea Severity and Risk of Atrial Fibrillation: The VARIOSA-AF Study. JACC Clin Electrophysiol. 2019 Jun;5(6):692-701. doi: 10.1016/j.jacep.2019.03.005. Epub 2019 May 1. PMID 31221356
- [Background] Oakes RS, Badger TJ, Kholmovski EG, Akoum N, Burgon NS, Fish EN, Blauer JJ, Rao SN, DiBella EV, Segerson NM, Daccarett M, Windfelder J, McGann CJ, Parker D, MacLeod RS, Marrouche NF. Detection and quantification of left atrial structural remodeling with delayed-enhancement magnetic resonance imaging in patients with atrial fibrillation. Circulation. 2009 Apr 7;119(13):1758-67. doi: 10.1161/CIRCULATIONAHA.108.811877. Epub 2009 Mar 23. PMID 19307477
- [Background] Marrouche NF, Wilber D, Hindricks G, Jais P, Akoum N, Marchlinski F, Kholmovski E, Burgon N, Hu N, Mont L, Deneke T, Duytschaever M, Neumann T, Mansour M, Mahnkopf C, Herweg B, Daoud E, Wissner E, Bansmann P, Brachmann J. Association of atrial tissue fibrosis identified by delayed enhancement MRI and atrial fibrillation catheter ablation: the DECAAF study. JAMA. 2014 Feb 5;311(5):498-506. doi: 10.1001/jama.2014.3. PMID 24496537
- [Background] Gal P, Marrouche NF. Magnetic resonance imaging of atrial fibrosis: redefining atrial fibrillation to a syndrome. Eur Heart J. 2017 Jan 1;38(1):14-19. doi: 10.1093/eurheartj/ehv514. Epub 2015 Sep 25. PMID 26409008
- [Background] King JB, Azadani PN, Suksaranjit P, Bress AP, Witt DM, Han FT, Chelu MG, Silver MA, Biskupiak J, Wilson BD, Morris AK, Kholmovski EG, Marrouche N. Left Atrial Fibrosis and Risk of Cerebrovascular and Cardiovascular Events in Patients With Atrial Fibrillation. J Am Coll Cardiol. 2017 Sep 12;70(11):1311-1321. doi: 10.1016/j.jacc.2017.07.758. PMID 28882227
- [Background] Otto ME, Belohlavek M, Romero-Corral A, Gami AS, Gilman G, Svatikova A, Amin RS, Lopez-Jimenez F, Khandheria BK, Somers VK. Comparison of cardiac structural and functional changes in obese otherwise healthy adults with versus without obstructive sleep apnea. Am J Cardiol. 2007 May 1;99(9):1298-302. doi: 10.1016/j.amjcard.2006.12.052. Epub 2007 Mar 20. PMID 17478161
- [Background] Dimitri H, Ng M, Brooks AG, Kuklik P, Stiles MK, Lau DH, Antic N, Thornton A, Saint DA, McEvoy D, Antic R, Kalman JM, Sanders P. Atrial remodeling in obstructive sleep apnea: implications for atrial fibrillation. Heart Rhythm. 2012 Mar;9(3):321-7. doi: 10.1016/j.hrthm.2011.10.017. Epub 2011 Oct 19. PMID 22016075
- [Background] Anter E, Di Biase L, Contreras-Valdes FM, Gianni C, Mohanty S, Tschabrunn CM, Viles-Gonzalez JF, Leshem E, Buxton AE, Kulbak G, Halaby RN, Zimetbaum PJ, Waks JW, Thomas RJ, Natale A, Josephson ME. Atrial Substrate and Triggers of Paroxysmal Atrial Fibrillation in Patients With Obstructive Sleep Apnea. Circ Arrhythm Electrophysiol. 2017 Nov;10(11):e005407. doi: 10.1161/CIRCEP.117.005407. PMID 29133380
- [Background] Iwasaki YK, Kato T, Xiong F, Shi YF, Naud P, Maguy A, Mizuno K, Tardif JC, Comtois P, Nattel S. Atrial fibrillation promotion with long-term repetitive obstructive sleep apnea in a rat model. J Am Coll Cardiol. 2014 Nov 11;64(19):2013-23. doi: 10.1016/j.jacc.2014.05.077. Epub 2014 Nov 3. PMID 25440097